CLINICAL TRIAL: NCT05760261
Title: A Phase 1, Open-Label Study in Healthy Participants Aged 18 to 65 Years to Investigate the CYP3A4 Induction Potential of GSK3882347
Brief Title: Drug Interaction Assessment of GSK3882347 in Healthy Participants Aged 18 to 65 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213252
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Urinary Tract Infections
Keywords: Drug-drug interaction; Cytochrome P450 3A4 (CYP3A4); 1-hydroxymidazolam; Hormonal contraceptive agent
MeSH Terms: conditions — Urinary Tract Infections | interventions — Midazolam

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GSK3882347 and MDZ (Experimental): Period 1: Participants will receive MDZ on Day 1. Period 2: Participants will receive 14-days of repeat dosing of GSK3882347 Followed by one dose of MDZ co-administered with GSK3882347 on Day 15.
  Interventions: Drug: Midazolam; Drug: GSK3882347

INTERVENTIONS:
Drug: Midazolam — Midazolam will be administered.
Drug: GSK3882347 — GSK3882347 will be administered.

SUMMARY:
The objective of this study is to determine the magnitude and clinical relevance of a potential drug-drug interaction of GSK3882347 with midazolam (MDZ) in healthy participants. This study assesses the effect of GSK3882347 as an inducer of Cytochrome P450 3A4 (CYP3A4) using MDZ, a sensitive substrate of hepatic and intestinal CYP3A4. The study will investigate MDZ pharmacokinetic (PK) effect in two dosing periods:

Period 1: A single dose of MDZ Period 2: 14-days of once daily repeat dosing of GSK3882347 followed by single dose of MDZ co-administered with GSK3882347 on Day 15 (14-days has been selected as this duration is required in order to maximize any potential CYP3A4 enzyme induction).

ELIGIBILITY:
Inclusion criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. A participant with a clinical abnormality or laboratory parameter(s) not specifically listed in the exclusion or exclusion criteria that is outside the reference range for the population being studied may be included only if the investigator, in consultation with the Medical Monitor (if required), agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight at least 50.0 kilogram (kg) (110 pound [lbs.]) for males and 45.0 kg (99 lbs.) for females; and body mass index (BMI) within the range 18.5 - 32.0 kg per meter square (kg/m^2) (inclusive).
* Male participants are eligible to participate if they agree to the following during the study intervention Period and for at least 3 days, after the last dose of study intervention:

  * Refrain from donating fresh unwashed semen

Plus, either:

• Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

OR

• Must agree to use contraception/barrier.

* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

  * Is a woman of non-childbearing potential (WONCBP) . OR
  * Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, with a failure rate of lesser than (<) 1 percent (%).
* A WOCBP must have a negative highly sensitive pregnancy test [urine or serum] as required by local regulations) within 24h before the first dose of study intervention.
* The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).

Exclusion Criteria:

* History or presence of significant cardiovascular, respiratory, hepatic, renal, urological, gastrointestinal, metabolic, endocrinological, hematological, immunologic, dermatologic, neurological or psychiatric disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data or in the opinion of the investigator places the participants at unacceptable risk or would make adhering to study procedures for the duration of the study difficult. Participants who have had a gastric bypass or a cholecystectomy are excluded from the study.
* Abnormal blood pressure, as determined by the investigator.
* Alanine transferase (ALT) value greater than (>)1.5 × upper limit of normal (ULN).
* Bilirubin value >1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* The participant has a current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* The participant has congenital long QT syndrome or known prolongation of the corrected QT (QTc) interval.
* The participant has any history of heart failure.
* The participant has a family history of QT prolongation or sudden death.
* The participant has any current or previous a history of episodes of symptomatic bradycardia or bradyarrhythmia.
* The participant has a QTc >450 millisecond (msec). Note: The QTc is the QT interval corrected for heart rate according to Fridericia formula, machine, or manual overread.

  11. The participant has anuria, oliguria, or impairment of renal function (GFR by Modification of diet in renal disease [MDRD] <90 milliliter per minute per 1.73 meter square [mL/min/1.73m^2] or serum creatinine > ULN or urine albumin-creatinine ratio [ACR] of ≥300 milligram per gram [mg/g] at screening).
* The participant must agree to and adhere to the concomitant therapy (including nondrug therapies) restrictions from the Screening Visit through to the end of the end of the study (including telephone visit).
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 56 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 30 days or 5 half-lives, whichever is longer, before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research.
* Current enrolment or past participation in this clinical study.
* Positive human immunodeficiency virus (HIV) antibody test.
* Presence of Hepatitis B surface antigen (HbsAg) at screening or within 3 months prior to first dose of study intervention.
* Hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* A positive confirmation of Coronavirus disease 2019 (COVID-19) infection, or high clinical index of suspicion for COVID-19.
* The participant, in the judgment of the investigator, would not be able or willing to comply with the protocol or complete the study.
* Regular alcohol consumption within 6 months prior to the study. An average weekly intake of >14 units for males or females. One unit is equivalent to approximately to 8 g of alcohol: a half-pint (approximately [~]240 mL) of beer, one glass (125 mL) of wine or one (25 mL) measure of spirits.
* Positive smoke breathalyzer indicative of smoking history at screening and each in-house admission to the clinical research unit or regular use of tobacco or nicotine-containing products (i.e., nicotine patches or vaporizing devices) within 3 months prior to screening.
* Regular use of combustible tobacco products, and non-combustible nicotine delivery systems, inclusive of cigarettes, cigars, pipes, and materials used to "vape".
* Any history of substance abuse or a positive urine test for drugs of abuse/ alcohol breath screen at screening or admission.
* Known hypersensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Contraindication for MDZ (i.e., Hypersensitivity to the active substance, benzodiazepines or to any of the excipients, myasthenia gravis, respiratory insufficiency, sleep apnea syndrome, severe hepatic impairment).
* Use of any products intended to treat medical conditions that are not approved by the governing health authority in a given country or region (for example, herbal medicine, health supplements, traditional medicine, homeopathic remedies, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Period 1: Area under the curve from time zero to 24 hours (AUC [0-24]) for plasma concentration of MDZ | Up to 24 hours
Period 1: AUC (0-24) for plasma concentration of 1-hydroxy-MDZ | Up to 24 hours
Period 2: AUC (0-24) for plasma concentration of MDZ | Up to 24 hours
Period 2: AUC (0-24) for plasma concentration of 1-hydroxy-MDZ | Up to 24 hours
Period 1: AUC from time zero to last time of quantifiable concentration (AUC [0-tau]) for plasma concentration of MDZ | Up to Day 2
Period 1: AUC (0-tau) for plasma concentration of 1-hydroxy-MDZ | Up to Day 2
Period 2: AUC (0-tau) for plasma concentration of MDZ | Up to Day 15
Period 2: AUC (0-tau) for plasma concentration of 1-hydroxy-MDZ | Up to Day 15
Period 1: AUC from time zero extrapolated to infinite time (AUC [0-inf]) for plasma concentration of MDZ | Up to Day 2
Period 1: AUC (0-inf) for plasma concentration of 1-hydroxy-MDZ | Up to Day 2
Period 2: AUC (0-inf) for plasma concentration of MDZ | Up to Day 15
Period 2: AUC (0-inf) for plasma concentration of 1-hydroxy-MDZ | Up to Day 15
Period 1: Maximum plasma concentration (Cmax) of MDZ | Up to Day 2
Period 1: Cmax of 1-hydroxy-MDZ | Up to Day 2
Period 2: Cmax of MDZ | Up to Day 15
Period 2: Cmax of 1-hydroxy-MDZ | Up to Day 15
Period 1: Time to Cmax (Tmax) of MDZ | Up to Day 2
Period 1: Tmax of 1-hydroxy-MDZ | Up to Day 2
Period 2: Tmax of MDZ | Up to Day 15
Period 2: Tmax of 1-hydroxy-MDZ | Up to Day 15
Period 1: Time lag before observation of measurable concentrations (Tlag) of MDZ | Up to Day 2
Period 1: Tlag of 1-hydroxy-MDZ | Up to Day 2
Period 2: Tlag of MDZ | Up to Day 15
Period 2: Tlag of 1-hydroxy-MDZ | Up to Day 15
Period 1: Time to half-life (T1/2) of MDZ | Up to Day 2
Period 1: T1/2 of 1-hydroxy-MDZ | Up to Day 2
Period 2: T1/2 of MDZ | Up to Day 15
Period 2: T1/2 of 1-hydroxy-MDZ | Up to Day 15

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 15
Number of participants with clinically significant changes in hematology laboratory values | Up to Day 15
Number of participants with clinically significant changes in chemistry laboratory values | Up to Day 15
Number of participants with clinically significant changes in urinalysis laboratory values | Up to Day 15
Number of participants with clinically significant changes in vital sign values | Up to Day 15
Number of participants with clinically significant changes in 12-lead electrocardiogram (ECG) readings | Up to Day 15
AUC (0-24) for plasma concentration of GSK3882347 | Up to 24 hours
Plasma concentrations over the dosing interval tau (Ctau) of GSK3882347 | Up to Day 15
Oral clearance (CL/F) of GSK3882347 | Up to Day 15
Volume of distribution/ Bioavailability (Vd/F) of GSK3882347 | Up to Day 15
Mean residence time (MRT) of GSK3882347 | Up to Day 15
AUC(0-inf) for single dose of GSK3882347 | Up to Day 2
Cmax for single dose of GSK3882347 | Up to Day 2
AUC(0-tau) for repeat dose of GSK3882347 | Up to Day 15
Cmax for repeat dose of GSK3882347 | Up to Day 15
Accumulation ratio (Ro) using AUC (0-tau) for repeat dose of GSK3882347 | Up to Day 15
Time invariance using AUC(0-tau) (repeat dose) of GSK3882347 | Up to Day 15
Time invariance using AUC(0-inf) (single dose) of GSK3882347 | Up to Day 2
Achievement of steady state of GSK3882347 | Up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/